CLINICAL TRIAL: NCT00612872
Title: Evaluation of [123I]CLINDE and SPECT as a Marker of Inflammation in Subjects With Parkinson Disease or Alzheimer Disease and in Healthy Subjects
Brief Title: Evaluation of [123I]CLINDE and SPECT as a Marker of Inflammation in Subjects With PD or AD and in Healthy Subjects
Acronym: CLINDE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Results did not show reason to continue with study.
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CLINDE 001; IND 100,863 (Other: IND Number)
Record Dates: First submitted 2008-01-16; First posted 2008-02-12 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease; Alzheimer Disease; Healthy Controls; Multiple Sclerosis
MeSH Terms: conditions — Parkinson Disease; Alzheimer Disease; Multiple Sclerosis | interventions — 6-chloro-2-(4'-iodophenyl)-3-(N,N-diethyl)imidazo(1,2-a)pyridine-3-acetamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assess [123-I]CLINDE and brain imaging (Experimental): Subjects will be injected with up to 5 mCi and not to exceed 5.5 (not >10% of 5 mCi limit) of 123-I CLINDE followed by serial SPECT imaging.
  Interventions: Drug: [123I]CLINDE

INTERVENTIONS:
Drug: [123I]CLINDE — Subjects will be injected with up to 5 mCi and not to exceed 5.5 (not >10% of 5 mCi limit) of 123-I CLINDE followed by serial SPECT imaging.

SUMMARY:
To assess the dynamic uptake and washout of 123-I CLINDE, a potential imaging biomarker for inflammatory changes in brain, using single photon emission computed tomography (SPECT) in similarly aged healthy controls and subjects with Alzheimer (AD) or Parkinson disease (PD).

To perform blood metabolite characterization of 123-I CLINDE in healthy and subjects with AD or PD to determine the nature of metabolites in assessment of 123-I CLINDE as a single photon computed tomography (SPECT) brain imaging agent.

Evaluate the test/retest reproducibility of 123-I CLINDE, and SPECT in AD and PD subjects and healthy controls

DETAILED DESCRIPTION:
When microglia become activated they express peripheral benzodiazepine receptors (PBR) or binding sites on their mitochondrial membrane. PBRs are functionally and structurally distinct from central benzodiazepine receptors associated with y-aminiobutric acid (GABA)-regulated chloride channels. PBRs are found in abundance in peripheral organs and hematologic cells, but are present at only very low levels in the normal central nervous system (Banati, 2002). CLINDE is a phenylimidazopyridine and appears to bind selectively to the PBR. In the absence of excessive blood in the CNS an increase CLINDE binding to PBR is a potential marker of microglial activation in the CNS. The increase in CLINDE binding may be an indicator of the transition of microglia from a resting to an activated state. When labeled with 123-I and used as a SPECT radiotracer, CLINDE may serve as an in vivo marker of microglial activation in Alzheimer disease and Parkinson disease.

The 123-I radioactive tag offers distinct advantages for large-scale clinical imaging studies of anti-inflammatory targeted treatments as a marker of microglial activation and efficacy of therapeutic intervention. The half-life (13.1 h) of 123-I permits imaging in multiple subjects in a single research-dedicated imaging center, with multiple research subjects per day. This minimizes variability introduced in multi-center quantitative imaging trials where different cameras, image processing methods, and QA procedures all conspire to increase the variance imaging biomarkers. Using this model, our group pioneered a method to evaluate the loss of dopamine function in Parkinson's disease using a radioactive drug 123-I β-CIT which binds directly to dopamine nerve terminals.

The adaptation of imaging agents like 123-I CLINDE as a biomarker of microglial activation in neurodegenerative diseases requires human validation studies. Expanding upon our previous work with b-amyloid ligands (123I-IMPY, 123-I MNI-187) for AD and dopamine transporter ligands (123-I B-CIT, Altropane) for PD, we desire to develop and characterize 123-I CLINDE as a potential marker for microglial activation in association with neuronal damage that may be applicable to multiple neurodegenerative diseases. Ultimately a marker of microglial activation could be used for large-scale quantitative brain imaging trials in AD or PD, specifically to investigate the agent as an objective biomarker in treatments aimed at reducing inflammatory changes in these conditions. The significance of this work lies in applying state-of-art quantitative neuroimaging tools to develop a relevant biomarker in individuals with neurodegenerative diseases with the intention of using this efficiently in large clinical imaging trials.

ELIGIBILITY:
Inclusion Criteria:

Alzheimer's Subject Selection. Subjects who have a clinical diagnosis of mild to moderate Alzheimer's disease will be recruited for this study. The following criteria will be met for inclusion of AD subjects in this study:

* The participant is 50 years or older.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of probable Alzheimer's disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria.
* Mini-Mental Status Exam score < 25.
* Modified Hachinski Ischemia Scale score of ≤ 4.
* Geriatric Depression Scales (GDS) ≤ 10.
* For females, non-child bearing potential a negative urine or blood pregnancy test on day of 123-I CLINDE injection.

Parkinson's Subject Selection. Subjects who have a clinical diagnosis of mild to moderate Parkinson disease will be recruited for this study. The following criteria will be met for inclusion of PD subjects in this study:

* The participant is 30 years or older.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of Parkinson disease (at least two of the three cardinal symptoms: resting tremor, rigidity, bradykinesia).
* Geriatric Depression Scales (GDS) ≤ 10.
* Hoehn and Yahr ≤4.
* For females, non-child bearing potential a negative urine or blood pregnancy test on day of 123-I CLINDE injection.

Healthy Control Subject Selection. Healthy control subjects who have no neurological disease will be recruited for this study. The following criteria will be met for inclusion of healthy control subjects in this study:

* The participant is 30 years or older.
* Written informed consent is obtained.
* Negative history of neurological or psychiatric illness based on evaluation by a research physician.
* Mini-Mental Status Exam score ≥28.
* For females, non-child bearing potential a negative urine or blood pregnancy test on day of 123-I CLINDE injection.

Exclusion Criteria:

Alzheimer's subjects will be excluded from participation for the following reasons:

* The subject has a history of significant cerebrovascular disease.
* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Pregnancy
* Positive urine drug test.

Parkinson's subjects will be excluded from participation for the following reasons:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Pregnancy
* Positive urine drug test.

Healthy control subjects will be excluded from participation for the following reasons:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Pregnancy
* Positive urine drug test.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11-01 (Actual); Study Completion 2009-11-01 (Actual)

PRIMARY OUTCOMES:
To assess the dynamic uptake and washout of 123-I CLINDE, using single photon emission computed tomography (SPECT) in similarly aged healthy controls and subjects with Alzheimer (AD) or Parkinson disease (PD). | 6 mos

CONTACTS AND LOCATIONS:
Overall Officials: Danna L Jennings, M.D., Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- [Background] Aktas O, Ullrich O, Infante-Duarte C, Nitsch R, Zipp F. Neuronal damage in brain inflammation. Arch Neurol. 2007 Feb;64(2):185-9. doi: 10.1001/archneur.64.2.185. PMID 17296833
- [Background] Nomenclature and research case definitions for neurologic manifestations of human immunodeficiency virus-type 1 (HIV-1) infection. Report of a Working Group of the American Academy of Neurology AIDS Task Force. Neurology. 1991 Jun;41(6):778-85. doi: 10.1212/wnl.41.6.778. No abstract available. PMID 2046917
- See also: IND web page — http://www.indd.org